CLINICAL TRIAL: NCT04937452
Title: Dopaminergic Therapy for Frontotemporal Dementia Patients: an Interventional, Multi-site, Randomized, Double-blind, Placebo-controlled Study on the Efficacy and Safety of RTG Treatment in Patients with Behavioral FTD
Brief Title: Dopaminergic Therapy for Frontotemporal Dementia Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Collaborators: Alzheimer's Drug Discovery Foundation (Other)
Responsible Party: Principal Investigator, Giacomo Koch, Prof, I.R.C.C.S. Fondazione Santa Lucia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT 2019-002997-30
Record Dates: First submitted 2021-06-16; First posted 2021-06-24 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2022-07

CONDITIONS: Frontotemporal Dementia; Dementia; Aphasia, Primary Progressive; Pick Disease of the Brain; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Neurocognitive Disorders; Mental Disorders; Neurodegenerative Diseases; Frontotemporal Lobar Degeneration; TDP-43 Proteinopathies; Proteostasis Deficiencies; Metabolic Disease; Aphasia; Speech Disorders; Language Disorders; Communication Disorders; Neurobehavioral Manifestations; Neurologic Manifestations
Keywords: dopamine; frontal cortex; FTD; Rotigotine
MeSH Terms: conditions — Frontotemporal Dementia; Dementia; Aphasia, Primary Progressive; Pick Disease of the Brain; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Neurocognitive Disorders; Mental Disorders; Neurodegenerative Diseases; Frontotemporal Lobar Degeneration; TDP-43 Proteinopathies; Proteostasis Deficiencies; Metabolic Diseases; Aphasia; Speech Disorders; Language Disorders; Communication Disorders; Neurobehavioral Manifestations; Neurologic Manifestations | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Rotigotine 4 mg (Experimental): Rotigotine 4 mg/24 hours transdermal patch administration
  Interventions: Drug: Rotigotine 4Mg/24Hrs Patch
- Rotigotine 6 mg (Experimental): Rotigotine 6 mg/24 hours transdermal patch administration
  Interventions: Drug: Rotigotine 6Mg/24Hrs Patch
- Placebo (Placebo Comparator): Placebo transdermal patch administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rotigotine 4Mg/24Hrs Patch — Rotigotine 4 mg/24Hrs administration for 24 weeks
  Other Names: Neupro
  Arms: Rotigotine 4 mg
Drug: Rotigotine 6Mg/24Hrs Patch — Rotigotine 6 mg/24Hrs administration for 24 weeks
  Other Names: Neupro
  Arms: Rotigotine 6 mg
Drug: Placebo — Placebo administration for 24 weeks
  Arms: Placebo

SUMMARY:
This is a phase IIa 24-week randomized, double-blind, placebo-controlled study. The study is designed to evaluate the efficacy and safety of Rotigotine (RTG) transdermal administration at the dosage of 4 mg or 6 mg per day versus Placebo (PLC) in newly diagnosed behavioural Frontotemporal Dementia (bvFTD) patients. 75 patients with a diagnosis of probable bvFTD will be randomly allocated to the 3 treatment arms (RTG 4mg/day, RTG 6mg/day or PLC), with 25 patients per group. Clinical and neurophysiological measurements and brain metabolism via FDG-PET will be collected before and after drug administration.

DETAILED DESCRIPTION:
The current study has the ambition to provide the first-time evidence of the clinical impact, at cognitive and behavioral level, of a dopamine-based treatment in newly diagnosed bvFTD patients.

To evaluate the cognitive and behavioral effects of RTG administration, the investigators will employ a battery of tests assessing global cognition, executive functions, language and behavior.

The battery will include: Neuropsychiatric Inventory (NPI) and Frontal Behavioral Inventory (FBI) to evaluate behavior, Clinical Dementia Rating Scale-Frontotemporal Dementia Sum Of Boxes (CDR-FTD SOB) to evaluate global disease severity, Frontal Assessment Battery (FAB) to evaluate frontal functions, Screening for aphasia in Neurodegeneration (SAND) to evaluate language functions, Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) to evaluate activities of daily living, the Addenbrooke's Cognitive Examination Revised (ACE-R) to evaluate global cognition.

To evaluate changes in brain metabolism the investigators will perform 2 FDG-PET scans before starting the treatment and at the end of week 24.

Neurophysiological investigations will be performed to identify quantifiable biomarkers underlying the effects induced by dopamine agonist on the bvFTD brain. In particular, the investigators will use multimodal neurophysiological tools based on TMS-EMG and TMS-EEG. More specifically, different paired-pulse TMS protocols will be used to evaluate in vivo the activity of different intracortical circuits, such as short intracortical inhibition (SICI), reflecting GABA(A)-ergic neurotransmission; long intracortical inhibition (LICI), evaluating GABA(B)-ergic neurotransmission; short afferent inhibition (SAI) evaluating cholinergic neurotransmission and intermittent theta burst stimulation (iTBS) probing cortical plasticity mechanisms, such as long- term potentiation (LTP). The effects of these protocols will be evaluated by means of motor-evoked potentials, recordable with EMG. TMS-EEG will be used to measure the effects of RTG on frontal and parieto-temporal cortical activity, in terms of cortical excitability, oscillatory activity and connectivity. The investigators will evaluate the effects of the DA drug on brain activity and plasticity by analyzing MEPs and TEPs before and after the treatment. The investigators expect to find modulations in the high EEG frequencies (beta and gamma oscillatory activities) and/or in the indexes of cortical reactivity and plasticity (amplitude of TEPs and MEPs) that correlate with improvement in clinical assessment.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has a diagnosis of probable Frontotemporal dementia behavioural variant (bv-FTD) based on the International consensus clinical diagnostic criteria described by Rascovsky et al., 2011.
2. The patient is a man or a woman, aged from 40 to 80 years.
3. The patient has a Clinical Dementia Rating-FTD (CDR-FTD) total score of ≤2 at Screening.
4. The patient has not been treated with acetylcholinesterase inhibitor (AChEI), i.e., donepezil, galantamine, or rivastigmine, at the time of screening.
5. The patient is able to comply with the study procedures in the view of the investigator.
6. Evidence of frontotemporal hypometabolism at PET imaging.
7. Evidence of amyloid markers excluding Alzheimer's disease (cerebrospinal fluid Abeta/Tau dosages or amyloid PET imaging).
8. Signature and date of written ICF prior to entering in the study
9. Female patient must be neither pregnant nor breastfeeding. Women of childbearing potential should be willing to use contraception while receiving Rotigotine and for six months after its last assumption

Exclusion Criteria:

1. Significant neurodegenerative disorder of the central nervous system other than FTD e.g., Alzheimer's disease, Lewy body dementia, Parkinson's disease, multiple sclerosis, progressive supranuclear palsy, normal pressure hydrocephalus, Huntington's disease, any condition directly or indirectly caused by Transmissible Spongiform Encephalopathy (TSE), Creutzfeldt-Jakob Disease (CJD), variant Creutzfeldt-Jakob Disease (vCJD), or new variant Creutzfeldt-Jakob Disease (nvCJD)
2. Significant intracranial focal or vascular pathology seen on brain MRI scan within a maximum of 6 months before Baseline leading to a diagnosis other than probable FTD.
3. The patients has history of seizure (with the exception of febrile seizures in childhood).
4. Metal implants in the head (except dental), pacemaker, cochlear implants, or any other non-removable items that are contraindications to MR imaging.
5. Treatment currently or within 3 months before Baseline with any of the following medications: Typical and Atypical antipsychotics (i.e., Clozapine, Olanzapine); Antiepileptics drugs (i.e., Carbamazepine, Primidone, Pregabalin, Gabapentin); Antidepressants (i.e., Citalopram, Duolxetine, Paroxetine).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Frontal Assessment Battery (FAB) | 24 weeks
  Battery to evaluate executive functions. The scores range from 0-18 with a higher score meaning less cognitive impairment.

SECONDARY OUTCOMES:
Neuropsychiatric Inventory (NPI) scale | 24 weeks
  Battery to assess behavioral changes. The scores range from 0-144 with a higher score meaning more severe behavioural disturbances.
Frontal Behavioural Inventory (FBI) | 24 weeks
  Battery to assess behavioral changes. The scores range from 0-72 with a higher score meaning more severe behavioural disturbances.
Clinical Dementia Rating scale-Frontotemporal dementia Sum Of Boxes (CDR-FTDSOB) | 24 weeks
  Battery to evaluate global disease severity. The scores range from 0-24 with a higher score meaning higher disease severity.
Screening for aphasia in Neurodegeneration (SAND) scale | 24 weeks
  Battery to evaluate language functions. The scores range from 0-84 with a higher score meaning less severe language deficits.
Mini Mental State Examination (MMSE) | 24 weeks
  battery to evaluate global cognition. The scores range from 0-30 with a higher score meaning less cognitive impairment.
Addenbrooke's Cognitive Examination Revised (ACE-R) | 24 weeks
  battery to evaluate global cognition. The scores range from 0-100 with a higher score meaning less cognitive impairment.
Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) | 24 weeks
  battery to evaluate activities of daily living. The scores range from 0-78 with lower scores indicating more severe functional impairment.
CGIC questionnaire | 24 weeks
  questionnaire to evaluate clinically meaningful change
18F-FDG CT/PET | 24 weeks
  Change in brain glucose metabolism will be measured via FDG-PET
Long intracortical inhibition (LICI) | 24 weeks
  TMS protocol to evaluate GABA(B)ergic transmission
Short intracortical inhibition (SICI) | 24 weeks
  TMS protocol to evaluate GABA(B)ergic transmission
Short-Latency Afferent Inhibition (SAI) | 24 weeks
  TMS protocol to evaluate cholinergic transmission
Intermittent Theta Burst Stimulation (iTBS) | 24 weeks
  TMS protocol to evaluate cortical plasticity
TMS-EEG | 24 weeks
  power in beta-gamma band to evaluate prefrontal cortical oscillatory activity
Nature, frequency and severity of adverse events (AEs) | 24 weeks
  To assess the safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Koch, MD, Principal Investigator — Santa Lucia Foundation IRCCS; Martina Assogna, MD, Study Director — Santa Lucia Foundation IRCCS; Alessandro Martorana, MD, PhD, Study Chair — University of Tor Vergata
Locations (3):
- Italy (3):
  - Giacomo Koch, Rome, <None>
  - Department of Neurology, University of Brescia, Brescia
  - Santa Lucia Foundation, Rome

REFERENCES:
- [Derived] Koch G, Assogna M, Gadola Y, Alberici A, Di Lorenzo F, Bonni S, Borghi I, Cerulli Irelli E, Mencarelli L, Maiella M, Esposito R, Casula EP, Pezzopane V, D'Acunto A, Candeo F, Ferraresi M, Guerrera G, Battistini L, Premi E, Bracca V, Lucchini S, Bertagna F, Romano P, Ludovici A, Daniele A, Motta C, Ferrari C, Martorana A, Borroni B. Safety and efficacy of rotigotine in patients with frontotemporal dementia: a phase 2, double-blind, randomized, placebo-controlled, multicenter trial. Lancet Reg Health Eur. 2025 Aug 5;57:101409. doi: 10.1016/j.lanepe.2025.101409. eCollection 2025 Oct. PMID 40809903